CLINICAL TRIAL: NCT00512148
Title: An Open Label Multicenter Study of Augmentation Cystoplasty Using an Autologous Neo-Bladder Construct in Subjects With Neurogenic Bladder Following Spinal Cord Injury
Brief Title: Study of Autologous Neo-Bladder Construct in Subjects With Neurogenic Bladder Following Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 24 months follow up completed without substantial change to the profile.
Sponsor: Tengion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNG-CL004; NOTE: TENGION NO LONGER EXISTS (Other: NOTE: TENGION NO LONGER EXISTS FOLLOWING CHAPTER 7 BANKRUPTCY IN 2014. NO FURTHER INFORMATION IS AVAILABLE.)
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Note: Tengion no longer exists following Chapter 7 bankruptcy in 2014. No further information is available. No data are available to be reviewed or re-analyzed.
Masking Description: Note: Tengion no longer exists following Chapter 7 bankruptcy in 2014. No further information is available. No data are available to be reviewed or re-analyzed.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receipt of autologous neo-bladder construct consisting of a device regenerated in the laboratory from the patient's own muscle and urothelial cells
  Interventions: Device: Autologous neobladder construct

INTERVENTIONS:
Device: Autologous neobladder construct — augmentation cystoplasty with autologous neo-bladder construct

SUMMARY:
Subjects with neurogenic bladder secondary to spinal cord injury that is refractory to medical treatment and requires augmentation cystoplasty will be enrolled. The hypothesis is that augmentation cystoplasty using an autologous neo-bladder construct will reduce maximum detrusor pressure.

ELIGIBILITY:
Inclusion Criteria:

* subjects with neurogenic bladders secondary to spinal cord injury

Exclusion Criteria:

* prior augmentation procedures or urinary diversion
* recent urologic or intraperitoneal surgery or device implantation
* recent history of spinal cord injury of less than a year
* recent neurologic surgery
* requirement for concomitant urological surgical procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Sheth, MD, Study Director — Tengion, Inc
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 patients were recruited between September 2007 and October 2008. Patients were recruited from 4 academic centers across the US. 1 patient withdrew consent prior to bladder biopsy and is included in the safety analysis but not in the efficacy analysis. Due to recruitment challenges, only 6 patients were implanted.
Pre-assignment Details: This was an open label, single arm study.
Groups:
- Enterocystoplasty With the Neo-bladder Augment: Patients were enrolled who required enterocystoplasty (bladder augmentation). Patients in this study were augmented with with the Tengion neo-bladder augment. During this procedure the neo-bladder augment was surgically attached to the patient's existing bladder to enlarge its size.
Period: Primay Study Period
Arm/Group | Enterocystoplasty With the Neo-bladder Augment
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Long Term Follow Up Period
Arm/Group | Enterocystoplasty With the Neo-bladder Augment
Started | 6
Completed | 0 (6 patients are being followed in long term follow up)
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Enterocystoplasty With the Neo-bladder Augment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Detrusor Pressure From Baseline to 12 Months
Description: Detrusor pressure is measured using urodynamic testing, which involves inserting a catheter through the urethra and into the bladder and measuring the pressure in the bladder as it is filled with fluid. The primary outcome measure for this study was the change in the maximum pressure observed during bladder filling from baseline to 12 months. The goal of the therapy was to decrease pressure.
Time Frame: baseline and 12 months
Population: All patients with urodynamics measurement performed at baseline and month 12 were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: centimeters of water (cm H2O)
Groups:
- All Implanted: The number of subjects implanted with the neobladder augment
Arm/Group | All Implanted
Number analyzed (Participants) | 5
centimeters of water (cm H2O) | -17.0 [-61.4 to 27.4]

2. Primary Outcome: Overall Safety Profile - Number of Participants Experiencing an Adverse Event
Description: Clinical evaluation of adverse events experienced by patients enrolled in the trial.
Time Frame: through month 12
Population: This analysis was performed on the safety population. Patients undergoing screening and meeting inclusion/exclusion criteria were included in the safety population. Tengion no longer exists following Chapter 7 bankruptcy in 2014. No further data analysis will be made.
Measure: Number; unit: participants
Arm/Group | Enterocystoplasty With the Neo-bladder Augment
Number analyzed (Participants) | 7
participants | 7

3. Secondary Outcome: Urodynamic Measurements and Long Term Safety
Description: Safety results are summarized in the Adverse Events section of this listing.
Time Frame: month 12 through month 60
Population: Tengion no longer exists following Chapter 7 bankruptcy in 2014. No data were analyzed.
Groups:
- Patients Treated: Tengion no longer exists following Chapter 7 bankruptcy in 2014. No data were analyzed.
Arm/Group | Patients Treated
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: periodically within the first 12 months as well as during long term follow up out to 5 years.
Description: Adverse events are reported for 7 subjects who were enrolled in the study. One patient withdrew prior to bladder biopsy and is included in the safety population but not in the all implanted population used for efficacy analysis.
Groups:
- Safety Population: Patients who underwent screening procedures and met inclusion/exclusion criteria.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=7)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Post procedural urine leak (Injury, poisoning and procedural complications) | 3 (3)
Methicillin resistant Staphylococcus aureus test positive (Investigations) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=7)
Nausea (Gastrointestinal disorders) | 5 (11)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Pyrexia (General disorders) | 3 (4)
Edema peripheral (General disorders) | 2 (2)
Catheter site rash (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (18)
Bacteriuria (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (5)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (2)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (4)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (4)
Mental status changes (Psychiatric disorders) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator is free to individually communicate, orally present, or publish in scientific journals or other scholarly media the study information at the conclusion of the study without the prior approval of the sponsor provided that 1) the results of the study in its entirety have been publically disclosed by or with the consent of the sponsor 2)18 months after the conclusion of the study at all sites, whichever is first to occur.